CLINICAL TRIAL: NCT05003310
Title: Multipart Exploratory Study to Evaluate Splenic Nerve Stimulation in Patients With Rheumatoid Arthritis
Brief Title: ConsideRAte Study - Splenic Stimulation for RA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galvani Bioelectronics (Industry)
Collaborators: NAMSA (Other); Q2 Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GAL1040
Record Dates: First submitted 2021-07-05; First posted 2021-08-12 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Electrical stimulation; random allocation; inflammation; active implantable medical device; Laparoscopy; antirheumatic agents; autonomic nervous system; feasibility studies
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: Multicenter study with 4 periods. Period 1 is a randomized, controlled double-blind period where participants are assigned randomly to either active or sham stimulation. During the open-label Periods 2 through 4, participants are assigned treatment based on responses to treatments in the prior period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (7):
- Active Stimulation; Period 1 (Experimental): Active stimulation for 12 weeks
  Interventions: Device: Active Stimulation; Drug: Background Treatment
- Sham Stimulation; Period 1 (Sham Comparator): Sham stimulation for 12 weeks
  Interventions: Device: Sham Stimulation; Drug: Background Treatment
- Open label active stimulation, Period 2 (Experimental): Open label active stimulation for 12 additional weeks
  Interventions: Device: Active Stimulation; Drug: Background Treatment
- Open label RA Drug, Period 2 (Other): Open label drug treatment with baricitinib for 12 weeks
  Interventions: Drug: Baricitinib; Drug: Background Treatment
- RA drug combined with active stimulation, Period 3 (Experimental): Participants on baricitinib during Period 2 will have active stimulation added for 24 weeks
  Interventions: Device: Active Stimulation; Drug: Baricitinib; Drug: Background Treatment
- Active stimulation combined with RA drug, Period 3 (Experimental): Participants on active stimulation during Period 2 will have baricitinib added for 24 weeks
  Interventions: Device: Active Stimulation; Drug: Baricitinib; Drug: Background Treatment
- Long-term Follow-up, Period 4 (Other): Standard of care treatments with or without stimulation
  Interventions: Device: Active Stimulation; Drug: Background Treatment

INTERVENTIONS:
Device: Active Stimulation — Stimulation will be turned ON and applied during each day of the period.
  Arms: Active Stimulation; Period 1; Active stimulation combined with RA drug, Period 3; Long-term Follow-up, Period 4; Open label active stimulation, Period 2; RA drug combined with active stimulation, Period 3
Device: Sham Stimulation — Sham stimulation will be provided during the period
  Arms: Sham Stimulation; Period 1
Drug: Baricitinib — Baricitinib (2 mg) is administered daily during the period.
  Arms: Active stimulation combined with RA drug, Period 3; Open label RA Drug, Period 2; RA drug combined with active stimulation, Period 3
Drug: Background Treatment — Stable dose of standard background treatment (e.g., csDMARD therapy)

SUMMARY:
This study will evaluate the safety, tolerability, and effects of stimulating the splenic neurovascular bundle (NVB) with the Galvani System, which consists of a lead, implantable pulse generator, external components and accessories. The study will consist of 4 study periods, including a Randomized Control Trial period (Period 1), an Open Label period (Period 2), a Treat-to-target period (Period 3), and a Long-term Follow-up period (Period 4). Participants eligible for implant will have active rheumatoid arthritis (RA) and have an inadequate response or intolerance to at least two biologic Disease Modifying Anti-Rheumatic Drugs (DMARDs) or JAK inhibitors (JAKis). A sufficient number of participants will be enrolled so that approximately 28 participants will undergo device implantation.

DETAILED DESCRIPTION:
Participants with active rheumatoid arthritis (RA) who receive the implantable system will be randomly assigned to receive either active stimulation or sham-stimulation for 12 weeks (Period 1).

Following Period 1, all participants will enter an open label phase (Period 2) during which participants who responded to stimulation will continue on stimulation; whereas participants who received sham stimulation, or were stimulation non-responders, will receive a market-approved RA drug for 12 weeks.

At the end of Period 2, participants who respond to their Period 2 therapy but still exhibit signs and symptoms of RA will enter the Treat-to-target period (Period 3); others will proceed to Period 4 (Long-term Follow-up). During the Treat-to-Target period, participants will be treated with dual therapy (stimulation in combination with the market-approved RA drug) for up to 24 weeks.

Period 4 provides long term safety follow up for all study participants for a period of 5 years. Participants may receive stimulation in combination with other approved and standard of care therapies, subject to a favorable benefit-risk assessment in the judgement of the treating rheumatologist.

ELIGIBILITY:
Inclusion Criteria:

* RA of at least six months duration, per 2010 ACR/EULAR criteria
* Male or female participants, 22-75 years of age
* Active RA
* Inadequate Response to at least 2 biologic DMARDs and/or JAK-inhibitors (JAKis) including at least one TNF inhibitor
* Have an appropriate washout from previously used biological DMARDs or JAKi
* Receiving current treatment with standard dose(s) of conventional synthetic DMARD(s) or have documented history of failure due to ineffectiveness or intolerance

Exclusion Criteria:

* Inability to provide informed consent
* Significant psychiatric disease or substance abuse
* History of unilateral or bilateral vagotomy
* Active or latent tuberculosis
* Known infection with human immunodeficiency virus (HIV); current acute or chronic hepatitis B or hepatitis C; previous hepatitis B
* Positive SARS COV 2 PCR screening test for COVID-19 infection (at the point of screening for this study)
* Currently implanted electrically active medical devices (e.g., cardiac pacemakers, automatic implantable cardioverter-defibrillators)
* Previous splenectomy

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | Up through the end of Period 1 (Period 1 is up to 12 weeks duration)
  Adverse Events (AEs) may include clinically significant findings from Laboratory Safety Assessments (clinical chemistry and hematology), vital signs (blood pressure, heart rate, respiratory rate, and body temperature), and 12-Lead EKG
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | During Period 2 (Period 2 is up to 12 weeks in duration beyond Period 1)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | During Period 3 (Period 3 is up to 24 weeks in duration beyond Period 2)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | During Period 4 (Period 4 is up to 5 years in duration beyond Period 3)

SECONDARY OUTCOMES:
Change in the 28 Joint Disease Activity Score 28 - C reactive protein (DAS28-CRP) | Baseline to 12 weeks (Period 1)
Change in the level of Lipopolysaccharide (LPS)-inducible release of Tumor Necrosis Factor (TNFα) in whole blood assay | Baseline to 12 weeks (Period 1)
Change in the level of LPS-inducible release of TNFα in whole blood assay | Baseline to 24 weeks (Period 2)
Change in the level of LPS-inducible release of Interleukin 6 (IL-6) in whole blood assay | Baseline to 12 weeks (Period 1)
Change in the level of LPS-inducible release of Interleukin 6 (IL-6) in whole blood assay | Baseline to 24 weeks (Period 2)
Change in the level of LPS-inducible release of IL-8 in whole blood assay | Baseline to 12 weeks (Period 1)
Change in the level of LPS-inducible release of IL-8 in whole blood assay | Baseline to 24 weeks (Period 2)
Change in the level of LPS-inducible release of IL-17 in whole blood assay | Baseline to 12 weeks (Period 1)
Change in the level of LPS-inducible release of IL-17 in whole blood assay | Baseline to 24 weeks (Period 2)
Change in DAS28-CRP | Baseline to 24 weeks (Period 2)
Change in DAS28-CRP | Baseline to 36 weeks (Period 3)
Change in DAS28-CRP | Baseline to 48 weeks (Period 3)
Change in Health Assessment Questionnaire Disability Index (HAQ-DI) score | Baseline to 12 weeks (Period 1)
Change in HAQ-DI score | Baseline to 24 weeks (Period 2)
Change in HAQ-DI score | Baseline to 36 weeks (Period 3)
Change in HAQ-DI score | Baseline to 48 weeks (Period 3)
Change in Short Form 36 (SF-36) physical component score | Baseline to 12 weeks (Period 1)
Change in SF-36 physical component score | Baseline to 24 weeks (Period 2)
Change in SF-36 physical component score | Baseline to 36 weeks (Period 3)
Change in SF-36 physical component score | Baseline to 48 weeks (Period 3)
Change in SF-36 mental component score | Baseline to 12 weeks (Period 1)
Change in SF-36 mental component score | Baseline to 24 weeks (Period 2)
Change in SF-36 mental component score | Baseline to 36 weeks (Period 3)
Change in SF-36 mental component score | Baseline to 48 weeks (Period 3)
Change in SF-36 domain score | Baseline to 12 weeks (Period 1)
Change in SF-36 domain score | Baseline to 24 weeks (Period 2)
Change in SF-36 domain score | Baseline to 36 weeks (Period 3)
Change in SF-36 domain score | Baseline to 48 weeks (Period 3)
To evaluate the usability of the external Galvani System devices and accessories | Through 48 weeks
  Summarize feedback collected on a questionnaire pertaining to the use of the external Galvani System devices
To evaluate the participants' perception of therapy and sensation | Through 48 weeks
  A form is provided to participants at each visit after randomization to describe any sensations that may be associated with the Galvani System
Evaluate device performance as assessed by tabulation of device deficiencies | Through 48 weeks
Change in DAS28-CRP in participants who remain on active stimulation during Period 2 | week 12 to week 24
Incidence of participants who remain on active stimulation achieving DAS28-CRP score <2.6 at the end of Period 2 | Time Frame: Week 24
Change in DAS28-CRP in participants who are given Drug treatment with baricitinib during Period 2 | week 12 to week 24
Incidence of a change in DAS28-CRP greater than 1.2 units in participants who are given Drug treatment with baricitinib during Period 2 | week 12 to week 24
Incidence of participants who are given drug treatment with baricitinib achieving DAS28-CRP score <2.6 at the end of Period 2 | Week 24

CONTACTS AND LOCATIONS:
Locations (14):
- United States (12):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Medvin Research - Covina, Covina, California
  - Medvin Research - Whittier, Whittier, California
  - The Osteoporosis & Clinical Trials Center, Hagerstown, Maryland
  - NYU Langone, Brooklyn, New York
  - Oregon Health & Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Altoona, Pennsylvania
  - Arthritis & Rheumatology Institute, Allen, Texas
  - St. David's Healthcare, Austin, Texas
  - Tekton Research, Austin, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Southwest Rheumatology Research, Mesquite, Texas
- Netherlands (2):
  - Academic Medical Center (AMC) Dept of Rheumatology & Clinical Immunology, Amsterdam
  - Maxima Medical Center, MMC, Eindhoven